CLINICAL TRIAL: NCT05148026
Title: Regional Citrate Anticoagulation for Continuous Renal Replacement Therapy During Veno-venous ECMO: a Crossover Randomized Controlled Study
Brief Title: Regional Citrate Anticoagulation for RRT During V-V ECMO
Acronym: CRRT ECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Marco Giani, Research Collaborator, University of Milano Bicocca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3732
Record Dates: First submitted 2021-10-26; First posted 2021-12-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: ARDS, Human; Acute Kidney Injury
Keywords: Extracorporeal Membrane Oxygenation; Acute Kidney Injury; ARDS; Renal Replacement Therapy
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Kidney Injury | interventions — Heparin; Continuous Renal Replacement Therapy; Dialysis Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulation sequence 1 (UFH+ RCA) (Active Comparator): UFH+ RCA first
  Interventions: Drug: Unfractionated heparin first
- Anticoagulation sequence 2 (UFH) (Active Comparator): UFH first
  Interventions: Drug: Unfractionated heparin + RCA first

INTERVENTIONS:
Drug: Unfractionated heparin + RCA first — Patients are randomized to receive this sequence of anticoagulation regimens: UFH+RCA / UFH / UFH+RCA / UFH / UFH+RCA / UFH
  Other Names: Start with CVVHD, BF 100-120 ml/min, dialysate 2000 ml/h, RCA + systemic anticoagulation
  Arms: Anticoagulation sequence 2 (UFH)
Drug: Unfractionated heparin first — Patients are randomized to receive this sequence of anticoagulation regimens: UFH / UFH+RCA / UFH / UFH+RCA / UFH / UFH+RCA
  Other Names: Start with CVVHD, BF 200 ml/h, dialysate 2000 ml/h, systemic anticoagulation only
  Arms: Anticoagulation sequence 1 (UFH+ RCA)

SUMMARY:
Anticoagulation is an essential component of all extracorporeal therapies. Currently locoregional citrate anticoagulation is the recommended technique for continuous renal replacement therapy (CRRT).

However, low clearance of citrate restricts its use to blood flow up to 150 mL/min, preventing its use in ECMO.

Renal replacement therapy (RRT) is commonly provided to ECMO patients with AKI. In presence of systemic heparinization for ECMO, additional anticoagulation for the CRRT circuit (i.e. RCA) is usually not employed.

Nevertheless, thrombosis occurs more frequently in the CRRT circuit than the oxygenator because of the slower blood flow.

The aim of this prospective, cross-over study is to assess, in patients undergoing CRRT during veno-venous ECMO (vv-ECMO), the efficacy and safety of adding regional citrate anticoagulation (RCA) for CRRT circuit anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in ICU
* V-V ECMO support for acute respiratory failure
* CRRT therapy for acute kidney injury

Exclusion Criteria:

* Pregnancy
* Pre-existing coagulation disorders
* Contraindication to heparin or citrate anticoagulation
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of CRRT circuit clotting according to anticoagulation regimen | According to the manufacturer recommendation elective RRT circuit replacement will be performed after 72 hours of circuit life.
  Rate of clotting in the intervention group (RCA+UFH) vs controls (UFH). I.e. : did the circuit clot in its 72h life?

SECONDARY OUTCOMES:
CRRT circuit "survival" analysis | According to the manufacturer recommendation elective RRT circuit replacement will be performed after 72 hours of circuit life.
  "Circuit life" of RRT circuits in the intervention group (RCA+UFH) vs controls (UFH), comparison between groups will be performed as time to event(clotting) by log-rank test and described by the kaplan meier approach. Circuit replacement for other reasons (e.g. transfer to radiology to undergo a CT scan) will be right censored
Comparison of platelets count, D-dimers, fibrinogen | 72 hours for each circuit
  Comparison of lab values of blood sampled during intervention (RCA+UFH) vs control (UFH). Values will be compared as absolute value and as a difference compared to each circuit baseline
Incidence of citrate anticoagulation side-effects | 72 hours for each circuit
  Total to ionized calcium ratio (marker of citrate accumulation), rate of hypersodiemia and alkalosis will be compared between intervention (RCA+UFH) and control (UFH)
To evaluate the anticoagulation effects of UFH and RCA | 72 hours for each circuit
  TEG analysis of blood samples with UFH vs UFH+RCA effect will be compared. Specifically, TEG R-time will be compared in blood sampled from circuit anti-coagulated with RCA+UFH vs UFH only

CONTACTS AND LOCATIONS:
Locations (1):
- ASST MONZA-Rianimazione Generale, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zarbock A, Kullmar M, Kindgen-Milles D, Wempe C, Gerss J, Brandenburger T, Dimski T, Tyczynski B, Jahn M, Mulling N, Mehrlander M, Rosenberger P, Marx G, Simon TP, Jaschinski U, Deetjen P, Putensen C, Schewe JC, Kluge S, Jarczak D, Slowinski T, Bodenstein M, Meybohm P, Wirtz S, Moerer O, Kortgen A, Simon P, Bagshaw SM, Kellum JA, Meersch M; RICH Investigators and the Sepnet Trial Group. Effect of Regional Citrate Anticoagulation vs Systemic Heparin Anticoagulation During Continuous Kidney Replacement Therapy on Dialysis Filter Life Span and Mortality Among Critically Ill Patients With Acute Kidney Injury: A Randomized Clinical Trial. JAMA. 2020 Oct 27;324(16):1629-1639. doi: 10.1001/jama.2020.18618. PMID 33095849
- [Result] Giani M, Scaravilli V, Stefanini F, Valsecchi G, Rona R, Grasselli G, Bellani G, Pesenti AM, Foti G. Continuous Renal Replacement Therapy in Venovenous Extracorporeal Membrane Oxygenation: A Retrospective Study on Regional Citrate Anticoagulation. ASAIO J. 2020 Mar;66(3):332-338. doi: 10.1097/MAT.0000000000001003. PMID 31045918
- [Result] Shum HP, Kwan AM, Chan KC, Yan WW. The use of regional citrate anticoagulation continuous venovenous hemofiltration in extracorporeal membrane oxygenation. ASAIO J. 2014 Jul-Aug;60(4):413-8. doi: 10.1097/MAT.0000000000000085. PMID 24727536
- [Result] Schilder L, Nurmohamed SA, Bosch FH, Purmer IM, den Boer SS, Kleppe CG, Vervloet MG, Beishuizen A, Girbes AR, Ter Wee PM, Groeneveld AB; CASH study group. Citrate anticoagulation versus systemic heparinisation in continuous venovenous hemofiltration in critically ill patients with acute kidney injury: a multi-center randomized clinical trial. Crit Care. 2014 Aug 16;18(4):472. doi: 10.1186/s13054-014-0472-6. PMID 25128022
- [Result] Stucker F, Ponte B, Tataw J, Martin PY, Wozniak H, Pugin J, Saudan P. Efficacy and safety of citrate-based anticoagulation compared to heparin in patients with acute kidney injury requiring continuous renal replacement therapy: a randomized controlled trial. Crit Care. 2015 Mar 18;19(1):91. doi: 10.1186/s13054-015-0822-z. PMID 25881975